CLINICAL TRIAL: NCT00158756
Title: A Phase III, Partially Blind, Randomized Study to Evaluate the Immunogenicity, Safety and Reactogenicity of GlaxoSmithKline (GSK) Biologicals' Tritanrix™-HepB and GSK Biologicals Kft's DTPw-HBV Vaccines as Compared to Concomitant Administration of Commonwealth Serum Laboratory's (CSL's) DTPw (Triple Antigen™) and GSK Biologicals' HBV (Engerix™-B), When Co-administered With GSK Biologicals' Oral Live Attenuated Human Rotavirus (HRV) Vaccine, to Healthy Infants at 3, 4½ and 6 Months of Age, After a Birth Dose of Hepatitis B Vaccine.
Brief Title: Immune Response Post Pry Vaccination of 2 Formulations of DTPw-HBV Vaccine Given With Rotavirus Vaccine to Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 104021
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2017-07-12 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2017-04

CONDITIONS: Hepatitis B
Keywords: Diphtheria; Pertussis; Prophylaxis; Hepatitis B diseases; Tetanus
MeSH Terms: conditions — Hepatitis B; Diphtheria; Whooping Cough; Tetanus | interventions — RIX4414 vaccine

ARMS (5):
- Tritanrix™-HepB+Rotarix™ Group (Experimental): Subjects received 3 doses of Tritanrix™-HepB vaccine at 3, 4.5 and 6 months of age, intramuscularly into the right anterolateral thigh concomitantly with 2 oral doses of Rotarix™ vaccine at 3 and 4.5 months of age.
  Interventions: Biological: Tritanrix™-HepB; Biological: Rotarix™
- Tritanrix™-HepB+Placebo Group (Experimental): Subjects received 3 doses of Tritanrix™-HepB vaccine at 3, 4.5 and 6 months of age, intramuscularly into the right anterolateral thigh concomitantly with 2 oral doses of Placebo for Rotarix™ vaccine at 3 and 4.5 months of age.
  Interventions: Biological: Tritanrix™-HepB; Drug: Placebo
- Zilbrix™+Rotarix™ Group (Active Comparator): Subjects received 3 doses of Zilbrix™ vaccine at 3, 4.5 and 6 months of age, intramuscularly into the right anterolateral thigh concomitantly with 2 oral doses of Rotarix™ vaccine at 3 and 4.5 months of age.
  Interventions: Biological: Rotarix™; Biological: Zilbrix™
- Zilbrix™+Placebo Group (Active Comparator): Subjects received 3 doses of Zilbrix™ vaccine at 3, 4.5 and 6 months of age, intramuscularly into the right anterolateral thigh concomitantly with 2 oral doses of Placebo for Rotarix™ vaccine at 3 and 4.5 months of age.
  Interventions: Biological: Zilbrix™; Drug: Placebo
- Triple Antigen™+Engerix™-B Group (Active Comparator): Subjects received 3 separate doses of Triple Antigen™ and Engerix™-B vaccines at 3, 4.5 and 6 months of age, intramuscularly into the left and right anterolateral thighs, respectively.
  Interventions: Biological: Triple Antigen™; Biological: Engerix™-B

INTERVENTIONS:
Biological: Tritanrix™-HepB — GSK Biologicals' combined diphtheria-tetanus-whole cell Bordetella pertussis -hepatitis B vaccine.
  Other Names: DTPw-HBV
  Arms: Tritanrix™-HepB+Placebo Group; Tritanrix™-HepB+Rotarix™ Group
Biological: Rotarix™ — GSK Biologicals' live attenuated human rotavirus vaccine
  Other Names: HRV vaccine
  Arms: Tritanrix™-HepB+Rotarix™ Group; Zilbrix™+Rotarix™ Group
Biological: Zilbrix™ — GSK Biologicals Kft's combined diphtheria-tetanus whole-cell B. pertussis-hepatitis B vaccine
  Other Names: DTPw-HBV Kft
  Arms: Zilbrix™+Placebo Group; Zilbrix™+Rotarix™ Group
Biological: Triple Antigen™ — Commonwealth Serum Laboratory's (CSL's) combined diphtheria-tetanus-whole cell B. pertussis vaccine.
  Other Names: DTPwcsl vaccine
  Arms: Triple Antigen™+Engerix™-B Group
Biological: Engerix™-B — GSK Biologicals' hepatitis B vaccine
  Other Names: HBV vaccine
  Arms: Triple Antigen™+Engerix™-B Group
Drug: Placebo — Placebo for the Rotarix™ vaccine
  Arms: Tritanrix™-HepB+Placebo Group; Zilbrix™+Placebo Group

SUMMARY:
To compare the two formulations of GSK Biologicals' DTPw-HBV vaccine to concomitant administration of CSL's DTPw vaccine and GSK Biologicals' HBV with respect to the antibody response to the diphtheria antigen after a three-dose primary vaccination course.

DETAILED DESCRIPTION:
Randomized study with five groups to receive one of the following vaccination regimens:

One of the two formulations of GSK Biologicals' DTPw-HBV + GSK Biologicals' HRV One of the two formulations of GSK Biologicals' DTPw-HBV + Placebo CSL's DTPw + GSK Biologicals' HBV

ELIGIBILITY:
Inclusion criteria:

* Subjects who the investigator believes that their parent/guardian can and will comply with the requirements of the protocol.
* Administration of one dose of hepatitis B vaccine at birth.
* A male or female between, and including, 11 and 17 weeks of age at the time of the first DTPw vaccination.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.

Exclusion criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs since birth.
* Planned administration/ administration of a vaccine not foreseen by the study protocol within 30 days before the first vaccine dose or planned administration during the study period with the exception of oral polio vaccine.
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination (no laboratory testing is required)
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.

Ages: 3 Weeks to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 308 (Actual)
Dates: Start 2005-09-12 (Actual); Primary Completion 2006-11-01 (Actual); Study Completion 2006-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- Russia (8):
  - GSK Investigational Site, Barnaul
  - GSK Investigational Site, Ivanteevka Moscow Region
  - GSK Investigational Site, Krasnoyarsk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Samara
  - GSK Investigational Site, Tomsk
  - GSK Investigational Site, Yekaterinburg

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 104021 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 104021 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 104021 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 104021 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 104021 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 104021 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Tritanrix-HepB+Rotarix Group: Subjects received 3 doses of Tritanrix-HepB vaccine at 3, 4.5 and 6 months of age, intramuscularly into the right anterolateral thigh concomitantly with 2 oral doses of Rotarix vaccine at 3 and 4.5 months of age.
- Tritanrix-HepB+Placebo Group: Subjects received 3 doses of Tritanrix-HepB vaccine at 3, 4.5 and 6 months of age, intramuscularly into the right anterolateral thigh concomitantly with 2 oral doses of Placebo for Rotarix vaccine at 3 and 4.5 months of age.
- Zilbrix+Rotarix Group: Subjects received 3 doses of Zilbrix vaccine at 3, 4.5 and 6 months of age, intramuscularly into the right anterolateral thigh concomitantly with 2 oral doses of Rotarix vaccine at 3 and 4.5 months of age.
- Zilbrix+Placebo Group: Subjects received 3 doses of Zilbrix vaccine at 3, 4.5 and 6 months of age, intramuscularly into the right anterolateral thigh concomitantly with 2 oral doses of Placebo for Rotarix vaccine at 3 and 4.5 months of age.
- Triple Antigen+Engerix-B Group: Subjects received 3 separate doses of Triple Antigen and Engerix-B vaccines at 3, 4.5 and 6 months of age, intramuscularly into the left and right anterolateral thighs, respectively.
Period: Overall Study
Arm/Group | Tritanrix-HepB+Rotarix Group | Tritanrix-HepB+Placebo Group | Zilbrix+Rotarix Group | Zilbrix+Placebo Group | Triple Antigen+Engerix-B Group
Started | 80 | 25 | 81 | 23 | 99
Completed | 75 | 25 | 73 | 22 | 96
Not Completed | 5 | 0 | 8 | 1 | 3
Not completed — Withdrawal by Subject | 5 | 0 | 6 | 1 | 3
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0
Not completed — Serious adverse event | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tritanrix-HepB+Rotarix Group | Tritanrix-HepB+Placebo Group | Zilbrix+Rotarix Group | Zilbrix+Placebo Group | Triple Antigen+Engerix-B Group | Total
Number analyzed (Participants) | 80 | 25 | 81 | 23 | 99 | 308
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 13.0 (1.70) | 13.4 (1.87) | 12.8 (1.39) | 12.8 (1.56) | 12.9 (1.33) | 12.93 (1.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 6 | 45 | 11 | 48 | 152
  Male | 38 | 19 | 36 | 12 | 51 | 156

OUTCOME MEASURES:

1. Primary Outcome: Seroprotection Status for Anti-diphteria (Anti-DT) Antibodies
Description: Seroprotection status (SP) defined vaccinated subjects with antibody concentrations greater than or equal to (≥) 0.1 international units per millitre (IU/mL) as assessed by the Enzyme-linked Immunosorbent Assay (ELISA) or ≥ 0.016 IU/mL by neautralization assay on Vero cells in subjects seronegative for ELISA.
Time Frame: At one month post dose 3 [PIII(M4)]
Population: The analysis were performed on the According-To-Protocol (ATP) cohort for immunogenicity included all evaluable subjects (i.e. those who met all eligibility criteria, complied with the procedures defined in the protocol, with no elimination criteria during the study) for whom data concerning immunogenicity measures were available.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Tritanrix-HepB+Rotarix Group | Tritanrix-HepB+Placebo Group | Zilbrix+Rotarix Group | Zilbrix+Placebo Group | Triple Antigen+Engerix-B Group
Number analyzed (Participants) | 68 | 20 | 62 | 17 | 87
IU/mL | 100 [94.7 to 100] | 100 [83.2 to 100] | 100 [94.2 to 100] | 100 [80.5 to 100] | 98.9 [93.8 to 100]

2. Secondary Outcome: Number of Seroprotected Subjects for Anti-DT Antibodies as Assessed by ELISA
Description: A seroprotected subject is a vaccinated subject with concentrations ≥ 0.1 IU/mL.
Time Frame: At one month post dose 3 [PIII(M4)]
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity included all evaluable subjects (i.e. those who met all eligibility criteria, complied with the procedures defined in the protocol, with no elimination criteria during the study) for whom data concerning immunogenicity measures were available.
Measure: Number; unit: Subjects
Arm/Group | Tritanrix-HepB+Rotarix Group | Tritanrix-HepB+Placebo Group | Zilbrix+Rotarix Group | Zilbrix+Placebo Group | Triple Antigen+Engerix-B Group
Number analyzed (Participants) | 68 | 20 | 62 | 17 | 87
Subjects | 65 | 17 | 60 | 17 | 85

3. Secondary Outcome: Number of Seroprotected Subjects for Anti-Hepatitis B (Anti-HBs) Antibodies
Description: A seroprotected subject was defined as a vaccinated subject with antibody concentrations ≥ 10 milli-international units per millilitre (mIU/mL).
Time Frame: At one most post dose 3 [PIII(M4)]
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | Tritanrix-HepB+Rotarix Group | Tritanrix-HepB+Placebo Group | Zilbrix+Rotarix Group | Zilbrix+Placebo Group | Triple Antigen+Engerix-B Group
Number analyzed (Participants) | 64 | 19 | 58 | 16 | 86
Subjects | 64 | 19 | 58 | 16 | 84

4. Secondary Outcome: Number of Seropositive Subjects With Anti-Bordetella Pertussis (Anti-BPT) Antibody Concentrations ≥ the Established Cut-off Values
Description: A seropositive subject was defined as a subject with Anti-BPT antibody concentrations ≥ 15 ELISA units per millilitre (EL.U/mL), as assessed by the Enzyme-Linked Immunosorbent Assay (ELISA).
Time Frame: At one month post dose 3 [PIII(M4)]
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | Tritanrix-HepB+Rotarix Group | Tritanrix-HepB+Placebo Group | Zilbrix+Rotarix Group | Zilbrix+Placebo Group | Triple Antigen+Engerix-B Group
Number analyzed (Participants) | 67 | 20 | 62 | 17 | 86
Subjects | 67 | 19 | 60 | 16 | 79

5. Secondary Outcome: Number of Subjects With Vaccine Response to BPT Antigen
Description: Vaccine response (VR) was defined as the appearance of antibodies in subjects seronegative at pre-vaccination and antibody concentrations ≥ the cut-off values post-vaccination in subjects who were seropositive at pre-vaccination.
Time Frame: At one month post dose 3 [PIII(M4)]
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | Tritanrix-HepB+Rotarix Group | Tritanrix-HepB+Placebo Group | Zilbrix+Rotarix Group | Zilbrix+Placebo Group | Triple Antigen+Engerix-B Group
Number analyzed (Participants) | 67 | 20 | 62 | 17 | 86
Subjects | 67 | 19 | 60 | 16 | 79

6. Secondary Outcome: Number of Seropositive Subjects With Anti-rotavirus (Anti-RV) Antibodies Above the Cut-off Values
Description: A seropositive subject was defined as a subject with anti-RV antibody concentrations ≥ 20 units per millilitre (U/mL).
Time Frame: At 2.5 months after dose 2 of Rotarix [PIII(M4)]
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | Tritanrix-HepB+Rotarix Group | Tritanrix-HepB+Placebo Group | Zilbrix+Rotarix Group | Zilbrix+Placebo Group
Number analyzed (Participants) | 60 | 17 | 55 | 17
Subjects | 42 | 0 | 41 | 0

7. Secondary Outcome: Number of Seroprotected Subjects for Anti-Tetanus (Anti-T) Antigen
Description: A seroprotected subject was defined as a vaccinated subject with anti-T antibody concentrations ≥ the cut-off value of 0.1 international units per millilitre (IU/mL).
Time Frame: At one month post dose 3 [PIII(M4)]
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | Tritanrix-HepB+Rotarix Group | Tritanrix-HepB+Placebo Group | Zilbrix+Rotarix Group | Zilbrix+Placebo Group | Triple Antigen+Engerix-B Group
Number analyzed (Participants) | 68 | 20 | 62 | 17 | 87
Subjects | 68 | 20 | 62 | 17 | 87

8. Secondary Outcome: Number of Seroprotected Subjects for Anti-Poliovirus Types 1, 2, 3 (Anti-Polio 1, 2, 3)
Description: A seroprotected subject was defined as a vaccinated subject with anti-Polio type 1,2 ,3 antibody titers ≥ 8
Time Frame: At one month post dose 3 [PIII(M4)]
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | Tritanrix-HepB+Rotarix Group | Tritanrix-HepB+Placebo Group | Zilbrix+Rotarix Group | Zilbrix+Placebo Group | Triple Antigen+Engerix-B Group
Number analyzed (Participants) | 58 | 18 | 57 | 15 | 79
Subjects
  Anti-Polio 1, [N=54,17,47,14,72] | 54 | 17 | 47 | 14 | 72
  Anti-Polio 2, [N=58,18,57,14,79] | 58 | 18 | 57 | 14 | 79
  Anti-Polio 3, [N=57,18,55,15,79] | 56 | 17 | 55 | 15 | 79

9. Secondary Outcome: Concentrations of Anti-HBs Antibodies
Description: Concentrations of anti-HB, antibodies, expressed as Geometric Mean Concentrations (GMCs), were measured in mIU/mL.
Time Frame: At one month post dose 3 [PIII(M4)]
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Tritanrix-HepB+Rotarix Group | Tritanrix-HepB+Placebo Group | Zilbrix+Rotarix Group | Zilbrix+Placebo Group | Triple Antigen+Engerix-B Group
Number analyzed (Participants) | 64 | 19 | 58 | 16 | 84
mIU/mL | 600.5 [473.1 to 762.3] | 732.7 [472.0 to 1137.3] | 789.8 [626.8 to 995.1] | 850.6 [527.7 to 1371.2] | 578.6 [442.3 to 757.0]

10. Secondary Outcome: Concentrations of Anti-DT Antibodies
Description: Concentrations of anti-DT antibodies, expressed as Geometric Mean Concentrations (GMCs), were measured in IU/mL.
Time Frame: At one month post dose 3 [PIII(M4)]
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Tritanrix-HepB+Rotarix Group | Tritanrix-HepB+Placebo Group | Zilbrix+Rotarix Group | Zilbrix+Placebo Group | Triple Antigen+Engerix-B Group
Number analyzed (Participants) | 68 | 20 | 62 | 17 | 87
IU/mL | 0.667 [0.517 to 0.862] | 0.545 [0.276 to 1.078] | 0.957 [0.725 to 1.262] | 0.906 [0.569 to 1.444] | 1.096 [0.869 to 1.381]

11. Secondary Outcome: Concentrations of Anti-T Antibodies
Description: Concentrations, expressed as Geometric Mean Concentrations (GMCs), were measured in international units per millillitre (IU/mL).
Time Frame: At one month post dose 3 [PIII(M4)]
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Tritanrix-HepB+Rotarix Group | Tritanrix-HepB+Placebo Group | Zilbrix+Rotarix Group | Zilbrix+Placebo Group | Triple Antigen+Engerix-B Group
Number analyzed (Participants) | 68 | 20 | 62 | 17 | 87
IU/mL | 3.138 [2.580 to 3.817] | 3.350 [2.173 to 5.164] | 3.737 [3.079 to 4.535] | 5.323 [3.411 to 8.306] | 3.319 [2.838 to 3.881]

12. Secondary Outcome: Concentrations of Anti-BPT Antibodies
Description: Concentrations, expressed as Geometric Mean Concentrations (GMCs), were measured in EL.U/mL.
Time Frame: At one month post dose 3 [PIII(M4)]
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Tritanrix-HepB+Rotarix Group | Tritanrix-HepB+Placebo Group | Zilbrix+Rotarix Group | Zilbrix+Placebo Group | Triple Antigen+Engerix-B Group
Number analyzed (Participants) | 67 | 20 | 62 | 17 | 86
EL.U/mL | 65.7 [57.9 to 74.5] | 50.8 [36.5 to 70.6] | 40.1 [33.8 to 47.5] | 37.2 [25.6 to 54.3] | 38.0 [32.5 to 44.4]

13. Secondary Outcome: Concentrations of Anti-RV Antibodies
Description: Concentrations, expressed as Geometric Mean Concentrations (GMCs), were measured in U/mL.
Time Frame: At 2.5 months post dose 2 of Rotarix [PIII(M4)]
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity included all evaluable subjects (i.e. those who met all eligibility criteria, complied with the procedures defined in the protocol, with no elimination criteria during the study) for whom data concerning immunogenicity measures were available.lysis
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | Tritanrix-HepB+Rotarix Group | Tritanrix-HepB+Placebo Group | Zilbrix+Rotarix Group | Zilbrix+Placebo Group
Number analyzed (Participants) | 60 | 17 | 55 | 17
U/mL | 96.4 [57.5 to 161.8] | 10.0 [10.0 to 10.0] | 93.1 [56.1 to 154.3] | 10.0 [10.0 to 10.0]

14. Secondary Outcome: Anti-Polio Type 1, 2, 3 Antibody Titers
Description: Anti-Polio type 1, 2 and 3 antibody titers were expressed as Geometric Mean Titers (GMTs).
Time Frame: At one month post dose 3 [PIII(M4)]
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Tritanrix-HepB+Rotarix Group | Tritanrix-HepB+Placebo Group | Zilbrix+Rotarix Group | Zilbrix+Placebo Group | Triple Antigen+Engerix-B Group
Number analyzed (Participants) | 58 | 18 | 57 | 15 | 79
Titers
  Anti-Polio 1, [N=54,17,47,14,72] | 900.7 [643.1 to 1261.5] | 1181.0 [604.4 to 2307.7] | 877.7 [612.3 to 1257.9] | 779.9 [391.3 to 1554.1] | 1155.0 [877.8 to 1519.7]
  Anti-Polio 2, [N=58,18,57,14,79] | 811.2 [655.3 to 1004.1] | 1024.0 [679.8 to 1542.2] | 774.2 [602.4 to 994.9] | 882.6 [538.2 to 1447.4] | 825.9 [661.7 to 1031.0]
  Anti-Polio 3, [N=57,18,55,15,79] | 326.6 [234.7 to 454.3] | 369.1 [163.6 to 832.8] | 313.3 [240.8 to 407.7] | 330.3 [185.4 to 588.4] | 351.3 [267.5 to 461.3]

15. Secondary Outcome: Number of Subjects With Solicited Local Symptoms
Description: Solicited local symptoms were pain, redness and swelling. Any = occurence of symptom regardless of intensity grade. Grade 3 pain = Significant pain at rest, pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling with a maximum diameter greater than 30 millimeters (mm).
Time Frame: During the 8-Day (Days 0-7) follow-up period
Population: The analysis was performed on the Total Vaccinated cohort which included all subjects with at least one vaccine administration documented and the symptom sheet filled in.
Measure: Number; unit: Subjects
Arm/Group | Tritanrix-HepB+Rotarix Group | Tritanrix-HepB+Placebo Group | Zilbrix+Rotarix Group | Zilbrix+Placebo Group | Triple Antigen+Engerix-B Group
Number analyzed (Participants) | 78 | 25 | 76 | 23 | 98
Subjects
  Any Pain, Dose 1 [N=78;25;76;23;98] | 40 | 13 | 46 | 14 | 51
  Grade 3 Pain, Dose 1 [N=78;25;76;23;98] | 6 | 0 | 8 | 4 | 13
  Any Redness, Dose 1 [N=78;25;76;23;98] | 49 | 15 | 54 | 17 | 61
  Grade 3 Redness, Dose 1 [N=78;25;76;23;98] | 8 | 1 | 6 | 1 | 8
  Any Swelling, Dose 1 [N=78;25;76;23;98] | 27 | 9 | 33 | 7 | 31
  Grade 3 Swelling, Dose 1 [N=78;25;76;23;98] | 7 | 1 | 4 | 3 | 8
  Any Pain, Dose 2 [N=76;25;75;22;96] | 31 | 11 | 36 | 11 | 43
  Grade 3 Pain, Dose 2 [N=76;25;75;22;96] | 3 | 0 | 3 | 1 | 8
  Any Redness, Dose 2 [N=76;25;75;22;96] | 48 | 16 | 58 | 15 | 61
  Grade 3 Redness, Dose 2 [N=76;25;75;22;96] | 3 | 0 | 3 | 0 | 4
  Any Swelling, Dose 2 [N=76;25;75;22;96] | 32 | 8 | 36 | 7 | 37
  Grade 3 Swelling, Dose 2 [N=76;25;75;22;96] | 1 | 1 | 3 | 0 | 6
  Any Pain, Dose 3 [N=76;25;75;22;96] | 35 | 8 | 34 | 10 | 41
  Grade 3 Pain, Dose 3 [N=76;25;75;22;96] | 3 | 1 | 5 | 1 | 5
  Any Redness, Dose 3 [N=76;25;75;22;96] | 48 | 16 | 53 | 15 | 57
  Grade 3 Redness, Dose 3 [N=76;25;75;22;96] | 2 | 1 | 3 | 0 | 11
  Any Swelling, Dose 3 [N=76;25;75;22;96] | 33 | 10 | 38 | 9 | 47
  Grade 3 Swelling, Dose 3 [N=76;25;75;22;96] | 2 | 1 | 4 | 2 | 4
  Any Pain, Across [N=78;25;76;23;98] | 51 | 17 | 58 | 18 | 62
  Grade 3 Pain, Across [N=78;25;76;23;98] | 9 | 1 | 11 | 6 | 22
  Any Redness, Across [N=78;25;76;23;98] | 60 | 20 | 65 | 20 | 77
  Grade 3 Redness, Across [N=78;25;76;23;98] | 10 | 2 | 11 | 1 | 18
  Any Swelling, Across [N=78;25;76;23;98] | 44 | 16 | 52 | 12 | 57
  Grade 3 Swelling, Across [N=78;25;76;23;98] | 9 | 2 | 8 | 4 | 16

16. Secondary Outcome: Number of Subjects With Any Solicited General Symptoms
Description: Assessed solicited general symptoms were diarrhea, drowsiness, fever [defined as rectal temperature equal to or above 38.0 degrees Celsius (°C)], irritability, loss of appetite [loss of appet.] and vomiting. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.5 °C. Related = symptom assessed by the investigator as related to the vaccination. Grade 3 loss of appetite = symptoms that prevents eating. Grade 3 diarrhea = ≥ 6 looser than normal stools per (/) day. Grade 3 vomiting = ≥ 3 episodes of vomiting/day.
Time Frame: During the 8-day period (Days 0-7) post-vaccination
Population: as for outcome 15
Measure: Number; unit: Subjects
Arm/Group | Tritanrix-HepB+Rotarix Group | Tritanrix-HepB+Placebo Group | Zilbrix+Rotarix Group | Zilbrix+Placebo Group | Triple Antigen+Engerix-B Group
Number analyzed (Participants) | 78 | 25 | 77 | 23 | 98
Subjects
  Any Diarrhea, Dose 1[N=78;25;77;23;98] | 6 | 0 | 5 | 1 | 1
  Grade 3 Diarrhea, Dose 1[N=78;25;77;23;98] | 0 | 0 | 0 | 0 | 0
  Related Diarrhea, Dose 1[N=78;25;77;23;98] | 4 | 0 | 4 | 0 | 1
  Any Drowsiness, Dose 1[N=78;25;77;23;98] | 50 | 16 | 52 | 15 | 56
  Grade 3 Drowsiness, Dose 1[N=78;25;77;23;98] | 1 | 1 | 1 | 1 | 6
  Related Drowsiness, Dose 1[N=78;25;77;23;98] | 42 | 9 | 49 | 13 | 48
  Any Fever, Dose 1[N=78;25;77;23;98] | 43 | 13 | 49 | 12 | 68
  Grade 3 Fever, Dose 1[N=78;25;77;23;98] | 1 | 0 | 1 | 1 | 2
  Related Fever, Dose 1[N=78;25;77;23;98] | 42 | 12 | 49 | 11 | 67
  Any Irritability, Dose 1[N=78;25;77;23;98] | 54 | 23 | 56 | 17 | 70
  Grade 3 Irritability, Dose 1[N=78;25;77;23;98] | 6 | 1 | 4 | 2 | 10
  Related Irritability, Dose 1[N=78;25;77;23;98] | 49 | 17 | 52 | 13 | 65
  Any Loss of appet., Dose 1[N=78;25;77;23;98] | 35 | 9 | 34 | 11 | 32
  Grade 3 Loss of appet., Dose 1[N=78;25;77;23;98] | 1 | 0 | 1 | 0 | 1
  Related Loss of appet., Dose 1[N=78;25;77;23;98] | 28 | 5 | 27 | 10 | 27
  Any Vomiting, Dose 1[N=78;25;77;23;98] | 9 | 1 | 7 | 1 | 11
  Grade 3 Vomiting, Dose 1[N=78;25;77;23;98] | 1 | 0 | 0 | 0 | 1
  Related Vomiting, Dose 1[N=78;25;77;23;98] | 4 | 0 | 5 | 0 | 8
  Any Diarrhea, Dose 2[N=76;25;75;22;96] | 1 | 0 | 3 | 2 | 3
  Grade 3 Diarrhea, Dose 2[N=76;25;75;22;96] | 0 | 0 | 0 | 0 | 0
  Related Diarrhea, Dose 2[N=76;25;75;22;96] | 0 | 0 | 2 | 2 | 2
  Any Drowsiness, Dose 2[N=76;25;75;22;96] | 29 | 9 | 32 | 11 | 41
  Grade 3 Drowsiness, Dose 2[N=76;25;75;22;96] | 1 | 0 | 0 | 0 | 2
  Related Drowsiness, Dose 2[N=76;25;75;22;96] | 26 | 7 | 31 | 9 | 35
  Any Fever, Dose 2[N=76;25;75;22;96] | 22 | 10 | 31 | 11 | 45
  Grade 3 Fever, Dose 2[N=76;25;75;22;96] | 0 | 0 | 1 | 0 | 1
  Related Fever, Dose 2[N=76;25;75;22;96] | 20 | 9 | 30 | 10 | 44
  Any Irritability, Dose 2[N=76;25;75;22;96] | 41 | 10 | 49 | 11 | 61
  Grade 3 Irritability, Dose 2[N=76;25;75;22;96] | 2 | 0 | 2 | 1 | 3
  Related Irritability, Dose 2[N=76;25;75;22;96] | 37 | 9 | 44 | 9 | 55
  Any Loss of appet., Dose 2[N=76;25;75;22;96] | 22 | 9 | 12 | 5 | 23
  Grade 3 Loss of appet., Dose 2[N=76;25;75;22;96] | 0 | 0 | 1 | 0 | 2
  Related Loss of appet., Dose 2[N=76;25;75;22;96] | 28 | 9 | 12 | 4 | 22
  Any Vomiting, Dose 2[N=76;25;75;22;96] | 3 | 0 | 4 | 0 | 8
  Grade 3 Vomiting, Dose 2[N=76;25;75;22;96] | 0 | 0 | 0 | 0 | 2
  Related Vomiting, Dose 2[N=76;25;75;22;96] | 2 | 0 | 3 | 0 | 6
  Any Diarrhea, Dose 3[N=76;25;73;22;96] | 1 | 0 | 0 | 0 | 0
  Grade 3 Diarrhea, Dose 3[N=76;25;73;22;96] | 0 | 0 | 0 | 0 | 0
  Related Diarrhea, Dose 3[N=76;25;73;22;96] | 0 | 0 | 0 | 0 | 0
  Any Drowsiness, Dose 3[N=76;25;73;22;96] | 25 | 13 | 26 | 13 | 36
  Grade 3 Drowsiness, Dose 3[N=76;25;73;22;96] | 1 | 0 | 1 | 0 | 0
  Related Drowsiness, Dose 3[N=76;25;73;22;96] | 22 | 7 | 24 | 11 | 33
  Any Fever, Dose 3[N=76;25;73;22;96] | 24 | 8 | 27 | 11 | 41
  Grade 3 Fever, Dose 3[N=76;25;73;22;96] | 0 | 2 | 1 | 0 | 1
  Related Fever, Dose 3[N=76;25;73;22;96] | 22 | 7 | 27 | 10 | 41
  Any Irritability, Dose 3[N=76;25;73;22;96] | 38 | 15 | 40 | 13 | 53
  Grade 3 Irritability, Dose 3[N=76;25;73;22;96] | 1 | 0 | 2 | 1 | 2
  Related Irritability, Dose 3[N=76;25;73;22;96] | 35 | 13 | 37 | 12 | 51
  Any Loss of appet., Dose 3[N=76;25;73;22;96] | 20 | 8 | 15 | 6 | 17
  Grade 3 Loss of appet., Dose 3[N=76;25;73;22;96] | 0 | 0 | 0 | 0 | 0
  Related Loss of appet., Dose 3[N=76;25;73;22;96] | 18 | 5 | 13 | 6 | 16
  Any Vomiting, Dose 3[N=76;25;73;22;96] | 3 | 1 | 2 | 0 | 7
  Grade 3 Vomiting, Dose 3[N=76;25;73;22;96] | 0 | 0 | 0 | 0 | 0
  Related Vomiting, Dose 3[N=76;25;73;22;96] | 3 | 1 | 2 | 0 | 5
  Any Diarrhea, Across[N=78;25;77;23;98] | 8 | 0 | 6 | 3 | 4
  Grade 3 Diarrhea, Across[N=78;25;77;23;98] | 0 | 0 | 0 | 0 | 0
  Related Diarrhea, Across[N=78;25;77;23;98] | 4 | 0 | 5 | 2 | 3
  Any Drowsiness, Across[N=78;25;77;23;98] | 58 | 19 | 54 | 19 | 68
  Grade 3 Drowsiness, Across[N=78;25;77;23;98] | 3 | 1 | 2 | 1 | 6
  Related Drowsiness, Across[N=78;25;77;23;98] | 50 | 13 | 52 | 18 | 62
  Any Fever, Across[N=78;25;77;23;98] | 54 | 20 | 59 | 17 | 80
  Grade 3 Fever, Across[N=78;25;77;23;98] | 1 | 0 | 3 | 1 | 4
  Related Fever, Across[N=78;25;77;23;98] | 53 | 18 | 59 | 15 | 78
  Any Irritability, Across[N=78;25;77;23;98] | 61 | 23 | 66 | 20 | 84
  Grade 3 Irritability, Across[N=78;25;77;23;98] | 8 | 1 | 7 | 3 | 12
  Related Irritability, Across[N=78;25;77;23;98] | 59 | 20 | 64 | 19 | 80
  Any Loss of appet., Across[N=78;25;77;23;98] | 43 | 14 | 39 | 14 | 48
  Grade 3 Loss of appet., Across[N=78;25;77;23;98] | 1 | 0 | 2 | 0 | 3
  Related Loss of appet., Across[N=78;25;77;23;98] | 39 | 13 | 34 | 12 | 45
  Any Vomiting, Across[N=78;25;77;23;98] | 12 | 2 | 12 | 1 | 20
  Grade 3 Vomiting, Across[N=78;25;77;23;98] | 1 | 0 | 0 | 0 | 3
  Related Vomiting, Across[N=78;25;77;23;98] | 7 | 1 | 10 | 0 | 14

17. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: Number of subjects with any unsolicited adverse events (AEs)
  An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 31-day (Days 0-30) follow-up period
Population: as for outcome 15
Measure: Number; unit: Subjects
Arm/Group | Tritanrix-HepB+Rotarix Group | Tritanrix-HepB+Placebo Group | Zilbrix+Rotarix Group | Zilbrix+Placebo Group | Triple Antigen+Engerix-B Group
Number analyzed (Participants) | 80 | 25 | 81 | 23 | 99
Subjects | 8 | 6 | 19 | 5 | 12

18. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From Month 0 to Month 4
Population: as for outcome 15
Measure: Number; unit: Subjects
Arm/Group | Tritanrix-HepB+Rotarix Group | Tritanrix-HepB+Placebo Group | Zilbrix+Rotarix Group | Zilbrix+Placebo Group | Triple Antigen+Engerix-B Group
Number analyzed (Participants) | 80 | 25 | 81 | 23 | 99
Subjects | 1 | 0 | 7 | 0 | 2

ADVERSE EVENTS:
Time Frame: Solicited local+general during the 8-day (Days 0-7) post vaccination; AEs within the 31-Day;SAEs up to study end at Month 4
Arm/Group | Tritanrix™-HepB+Rotarix™ Group | Tritanrix™-HepB+Placebo Group | Zilbrix™+Rotarix™ Group | Zilbrix™+Placebo Group | Triple Antigen™+Engerix™-B Group
Serious Adverse Events (participants affected / at risk) | 1/80 | 0/25 | 7/81 | 0/23 | 2/99
Other Adverse Events (participants affected / at risk) | 74/80 | 25/25 | 74/81 | 22/23 | 96/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tritanrix™-HepB+Rotarix™ Group (N=80) | Tritanrix™-HepB+Placebo Group (N=25) | Zilbrix™+Rotarix™ Group (N=81) | Zilbrix™+Placebo Group (N=23) | Triple Antigen™+Engerix™-B Group (N=99)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 3 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Injection site abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Intussusception (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Laryngotracheitis obstructive (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Overgrowth bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Tritanrix™-HepB+Rotarix™ Group (N=80) | Tritanrix™-HepB+Placebo Group (N=25) | Zilbrix™+Rotarix™ Group (N=81) | Zilbrix™+Placebo Group (N=23) | Triple Antigen™+Engerix™-B Group (N=99)
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 3 | 2 | 5
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 3 | 1 | 0 | 0
Pain (General disorders) | 51/78 | 17 | 58/76 | 18 | 62/98
Redness (General disorders) | 60/78 | 20 | 65/76 | 20 | 77/98
Swelling (General disorders) | 44/78 | 16 | 52/76 | 12 | 57/98
Diarrhea (General disorders) | 8/78 | 0 | 6/77 | 3 | 4/98
Drowsiness (General disorders) | 58/78 | 19 | 54/77 | 19 | 68/98
Fever (General disorders) | 54/78 | 20 | 59/77 | 17 | 80/98
Irritability (General disorders) | 61/78 | 23 | 66/77 | 20 | 84/98
Loss of appetite (General disorders) | 43/78 | 14 | 39/77 | 14 | 48/98
Vomiting (General disorders) | 12/78 | 2 | 12/77 | 1 | 20/98

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.